CLINICAL TRIAL: NCT01737736
Title: Validation of Neurokeeper's Algorithm on Patients Undergoing Carotid Endarterectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neurokeeper Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: NK-004
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing cartoid endarterectomy surgery
  Interventions: Device: Neurokeeper stroke detector

INTERVENTIONS:
Device: Neurokeeper stroke detector — Electrophisoloigcal monitoring

SUMMARY:
The primary objective of the study is to validate an EEG base algorithm system to detect and monitor changes in cerebral electrophysiological parameters as compared to clinical evaluation in patients undergoing Carotid Endarterectomy.

The secondary objectives is measure time from ICA clamping to algorithm asymmetry detection, time from clinical deterioration to algorithm asymmetry detection Thi study is a prospective, open label, single arm, self control, single center study.

This study will be conducted in 50 subjects according to the inclusions/exclusions criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Primary Carotid Endarterectomy under local anesthesia in symptomatic or asymptomatic patients.

Exclusion Criteria:

* General anesthesia
* Selective carotid artery shunting.
* Previous major hemispheric stroke.
* Any known major hemispheric lesion.
* Significant movement disorder.
* Local skull or skin affliction which prevents electrodes application.
* Any known condition which in the opinion of the investigator may interfere with the protocol implementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Carotid Endarterectomy
Sampling Method: Non-Probability Sample
Dates: Start 2013-06

PRIMARY OUTCOMES:
Neurological detrioration detection
  The primary objective of the study is to validate an EEG base algorithm system to detect and monitor changes in cerebral electrophysiological parameters as compared to clinical evaluation in patients undergoing Carotid Endarterectomy.

SECONDARY OUTCOMES:
Time from deterioration to detection
  The secondary objectives is measure time from ICA clamping to algorithm asymmetry detection, time from clinical deterioration to algorithm asymmetry detection

CONTACTS AND LOCATIONS:
Overall Officials: Moshe' Herskovitz, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel